CLINICAL TRIAL: NCT01521455
Title: A Phase I, Randomized, Open, Multi-center, Cross Over Study to Evaluate the Therapeutic Equivalence of Repeated Dose of HCP0910 250/50 μg to SeretideTM 250 DiskusTM in Asthmatic Patients
Brief Title: Therapeutic Equivalence Study of HCP0910 250/50 Mcg to Seretide 250 Diskus in Asthmatic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-FTOL-101
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCP0910 (Experimental): Fluticasone /salmeterol 250/50 combination capsule
  Interventions: Drug: HCP0910
- Seretide Diskus (Active Comparator): Seretide 250 Diskus
  Interventions: Drug: Seretide Diskus

INTERVENTIONS:
Drug: HCP0910 — 250/50, BID for 2 weeks
  Arms: HCP0910
Drug: Seretide Diskus — 250/50, BID for 2 weeks
  Arms: Seretide Diskus

SUMMARY:
The purpose of this study is to prove that HCP0910 is therapeutically equivalent to Seretide 250 Diskus when repeatedly dosed to Asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* age 20 ~ 75 inclusive
* Asthmatic diagnosis in more than 12 weeks from screening day
* Shows more than 12 % increase, and 200mL increase in FEV1 measure on Visit 2

Exclusion Criteria:

* Maintain controlled asthma for more than 4 weeks before screening
* Diagnosed as a severe asthmatic patients

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
mean change of morning predose FEV1 from baseline | day 14

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-mi Park, Ph.D, Study Director — Hanmi Pharmaceutical Co.
Locations (7):
- South Korea (7):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyunggi -do
  - Ajou University Hospital, Suwon, Gyunggi -do
  - Asan Medical Center, Seoul
  - Ewha Womans University Medical Center, Seoul
  - Hanyang University Hospital, Seoul
  - Samsung medical center, Seoul
  - Seoul National University, Seoul